CLINICAL TRIAL: NCT04226807
Title: Re-imagining the Postpartum Process: The Impact of Earlier Postpartum Contact on Attendance at Postpartum Visits and Maternal Wellbeing
Brief Title: Impact of Earlier Postpartum Contact on Postpartum Visit Compliance and Maternal Wellbeing
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low participation rate, study converted to a cohort study instead
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Talitha Bruney, MD, Assistant Professor of Obstetrics and Gynecology and Women's Health, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019-10372
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Postpartum Care
Keywords: Postpartum Care; Visit Attendance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Postpartum Contact (Experimental): Patient receive a phone call from research staff 2-3 weeks after giving birth in addition to routine postpartum visit
  Interventions: Other: Early Postpartum Phone Call
- Routine Postpartum Care (No Intervention): Patient receives routine postpartum visit only

INTERVENTIONS:
Other: Early Postpartum Phone Call — Participants receive a phone call 2-3 weeks after birth asking about overall wellbeing, screening for complications and postpartum depression and referring to lactation or WIC as needed.
  Arms: Early Postpartum Contact

SUMMARY:
The American College of Obstetricians and Gynecologists has recommended a paradigm shift in how postpartum care is instituted. They recommend that in addition to the normal 4-12 week postpartum visit, women receive contact with a provider within the first 3 weeks after giving birth. This RCT will randomize patients to routine care- 6-12 week postpartum visit alone- or enhanced care- routine care plus a phone call within the first 3 weeks postpartum. The patients will then be asked to complete a follow up survey at 6 months postpartum. The primary outcome measure would be rates of compliance with the 6-12 week postpartum visit. Secondary outcome measures will include breastfeeding rates, rates of postpartum depression, hospital readmission rates and met desire for contraception.

ELIGIBILITY:
Inclusion Criteria:

* Had a vaginal or cesarean delivery at the Jack D. Weiler Hospital
* Gestational age greater than or equal to 36 weeks
* Received prenatal care at the Comprehensive Family Care Center (CFCC) clinic

Exclusion Criteria:

- Fetal or neonatal death or demise

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-01-31 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Attendance at comprehensive postpartum care visit | 12 weeks postpartum
  Percentage of women attending comprehensive postpartum visit

SECONDARY OUTCOMES:
Breastfeeding rates at 6 months | 6 months postpartum
  Percentage of women exclusively breastfeeding, using combined breastfeeding and formula feeding or exclusively using formula.
Need for family planning met | 6 months postpartum
  Percentage of women who want to be using a birth control method who are using one
Social work referral | 6 months postpartum
  Percentage of women who attend a social work appointment
Repeat pregnancy within 6 months of delivery | 6 months postpartum
  Percentage of women with a positive pregnancy test since delivery
Readmission to the hospital | 6 months postpartum
  Percentage of women admitted to any Montefiore hospital
Acceptability of early visit | 6 months postpartum
  Percentage of women who were "Very Satisfied" or "Satisfied" with the early phone call

CONTACTS AND LOCATIONS:
Overall Officials: Talitha Bruney, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kassebaum NJ, Bertozzi-Villa A, Coggeshall MS, Shackelford KA, Steiner C, Heuton KR, Gonzalez-Medina D, Barber R, Huynh C, Dicker D, Templin T, Wolock TM, Ozgoren AA, Abd-Allah F, Abera SF, Abubakar I, Achoki T, Adelekan A, Ademi Z, Adou AK, Adsuar JC, Agardh EE, Akena D, Alasfoor D, Alemu ZA, Alfonso-Cristancho R, Alhabib S, Ali R, Al Kahbouri MJ, Alla F, Allen PJ, AlMazroa MA, Alsharif U, Alvarez E, Alvis-Guzman N, Amankwaa AA, Amare AT, Amini H, Ammar W, Antonio CA, Anwari P, Arnlov J, Arsenijevic VS, Artaman A, Asad MM, Asghar RJ, Assadi R, Atkins LS, Badawi A, Balakrishnan K, Basu A, Basu S, Beardsley J, Bedi N, Bekele T, Bell ML, Bernabe E, Beyene TJ, Bhutta Z, Bin Abdulhak A, Blore JD, Basara BB, Bose D, Breitborde N, Cardenas R, Castaneda-Orjuela CA, Castro RE, Catala-Lopez F, Cavlin A, Chang JC, Che X, Christophi CA, Chugh SS, Cirillo M, Colquhoun SM, Cooper LT, Cooper C, da Costa Leite I, Dandona L, Dandona R, Davis A, Dayama A, Degenhardt L, De Leo D, del Pozo-Cruz B, Deribe K, Dessalegn M, deVeber GA, Dharmaratne SD, Dilmen U, Ding EL, Dorrington RE, Driscoll TR, Ermakov SP, Esteghamati A, Faraon EJ, Farzadfar F, Felicio MM, Fereshtehnejad SM, de Lima GM, Forouzanfar MH, Franca EB, Gaffikin L, Gambashidze K, Gankpe FG, Garcia AC, Geleijnse JM, Gibney KB, Giroud M, Glaser EL, Goginashvili K, Gona P, Gonzalez-Castell D, Goto A, Gouda HN, Gugnani HC, Gupta R, Gupta R, Hafezi-Nejad N, Hamadeh RR, Hammami M, Hankey GJ, Harb HL, Havmoeller R, Hay SI, Pi IB, Hoek HW, Hosgood HD, Hoy DG, Husseini A, Idrisov BT, Innos K, Inoue M, Jacobsen KH, Jahangir E, Jee SH, Jensen PN, Jha V, Jiang G, Jonas JB, Juel K, Kabagambe EK, Kan H, Karam NE, Karch A, Karema CK, Kaul A, Kawakami N, Kazanjan K, Kazi DS, Kemp AH, Kengne AP, Kereselidze M, Khader YS, Khalifa SE, Khan EA, Khang YH, Knibbs L, Kokubo Y, Kosen S, Defo BK, Kulkarni C, Kulkarni VS, Kumar GA, Kumar K, Kumar RB, Kwan G, Lai T, Lalloo R, Lam H, Lansingh VC, Larsson A, Lee JT, Leigh J, Leinsalu M, Leung R, Li X, Li Y, Li Y, Liang J, Liang X, Lim SS, Lin HH, Lipshultz SE, Liu S, Liu Y, Lloyd BK, London SJ, Lotufo PA, Ma J, Ma S, Machado VM, Mainoo NK, Majdan M, Mapoma CC, Marcenes W, Marzan MB, Mason-Jones AJ, Mehndiratta MM, Mejia-Rodriguez F, Memish ZA, Mendoza W, Miller TR, Mills EJ, Mokdad AH, Mola GL, Monasta L, de la Cruz Monis J, Hernandez JC, Moore AR, Moradi-Lakeh M, Mori R, Mueller UO, Mukaigawara M, Naheed A, Naidoo KS, Nand D, Nangia V, Nash D, Nejjari C, Nelson RG, Neupane SP, Newton CR, Ng M, Nieuwenhuijsen MJ, Nisar MI, Nolte S, Norheim OF, Nyakarahuka L, Oh IH, Ohkubo T, Olusanya BO, Omer SB, Opio JN, Orisakwe OE, Pandian JD, Papachristou C, Park JH, Caicedo AJ, Patten SB, Paul VK, Pavlin BI, Pearce N, Pereira DM, Pesudovs K, Petzold M, Poenaru D, Polanczyk GV, Polinder S, Pope D, Pourmalek F, Qato D, Quistberg DA, Rafay A, Rahimi K, Rahimi-Movaghar V, ur Rahman S, Raju M, Rana SM, Refaat A, Ronfani L, Roy N, Pimienta TG, Sahraian MA, Salomon JA, Sampson U, Santos IS, Sawhney M, Sayinzoga F, Schneider IJ, Schumacher A, Schwebel DC, Seedat S, Sepanlou SG, Servan-Mori EE, Shakh-Nazarova M, Sheikhbahaei S, Shibuya K, Shin HH, Shiue I, Sigfusdottir ID, Silberberg DH, Silva AP, Singh JA, Skirbekk V, Sliwa K, Soshnikov SS, Sposato LA, Sreeramareddy CT, Stroumpoulis K, Sturua L, Sykes BL, Tabb KM, Talongwa RT, Tan F, Teixeira CM, Tenkorang EY, Terkawi AS, Thorne-Lyman AL, Tirschwell DL, Towbin JA, Tran BX, Tsilimbaris M, Uchendu US, Ukwaja KN, Undurraga EA, Uzun SB, Vallely AJ, van Gool CH, Vasankari TJ, Vavilala MS, Venketasubramanian N, Villalpando S, Violante FS, Vlassov VV, Vos T, Waller S, Wang H, Wang L, Wang X, Wang Y, Weichenthal S, Weiderpass E, Weintraub RG, Westerman R, Wilkinson JD, Woldeyohannes SM, Wong JQ, Wordofa MA, Xu G, Yang YC, Yano Y, Yentur GK, Yip P, Yonemoto N, Yoon SJ, Younis MZ, Yu C, Jin KY, El Sayed Zaki M, Zhao Y, Zheng Y, Zhou M, Zhu J, Zou XN, Lopez AD, Naghavi M, Murray CJ, Lozano R. Global, regional, and national levels and causes of maternal mortality during 1990-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet. 2014 Sep 13;384(9947):980-1004. doi: 10.1016/S0140-6736(14)60696-6. Epub 2014 May 2. PMID 24797575
- [Background] ACOG Committee Opinion No. 736: Optimizing Postpartum Care. Obstet Gynecol. 2018 May;131(5):e140-e150. doi: 10.1097/AOG.0000000000002633. PMID 29683911
- [Background] Wilcox A, Levi EE, Garrett JM. Predictors of Non-Attendance to the Postpartum Follow-up Visit. Matern Child Health J. 2016 Nov;20(Suppl 1):22-27. doi: 10.1007/s10995-016-2184-9. PMID 27562797
- [Background] Baldwin MK, Hart KD, Rodriguez MI. Predictors for follow-up among postpartum patients enrolled in a clinical trial. Contraception. 2018 Sep;98(3):228-231. doi: 10.1016/j.contraception.2018.04.016. Epub 2018 May 8. PMID 29750924
- [Background] Tsai PJ, Nakashima L, Yamamoto J, Ngo L, Kaneshiro B. Postpartum follow-up rates before and after the postpartum follow-up initiative at Queen Emma Clinic. Hawaii Med J. 2011 Mar;70(3):56-9. PMID 21365543
- [Background] Chen MJ, Hsia JK, Hou MY, Wilson MD, Creinin MD. Comparing Postpartum Visit Attendance with a Scheduled 2- to 3-Week or 6-Week Visit after Delivery. Am J Perinatol. 2019 Jul;36(9):936-942. doi: 10.1055/s-0038-1675623. Epub 2018 Nov 10. PMID 30414598
- [Background] Goulet L, D'Amour D, Pineault R. Type and timing of services following postnatal discharge: do they make a difference? Women Health. 2007;45(4):19-39. doi: 10.1300/J013v45n04_02. PMID 18032166
- See also: Healthcare Effectiveness Data and Information Set: Prenatal and Postpartum Care — https://www.ncqa.org/hedis/measures/prenatal-and-postpartum-care-ppc/